CLINICAL TRIAL: NCT06202859
Title: Respiratory Physiotherapy as a Tool to Increase the Number of Solid Organ Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vall d'Hebron Institute Research (Other)
Collaborators: Hospital Vall d'Hebron (Other); Germans Trias i Pujol Hospital (Other); Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Irene Bello, Professor, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIE-don study
Record Dates: First submitted 2023-10-23; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lung Transplant Failure
Keywords: respiratory physiotherapy; lung donor; improve lung donor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIE group (Experimental): * Manual techniques of secretion drainage
  * Two sequences separated for 1 min of 6 cycles each of MI-E(Cough Assist E70, Respironics Philips.
  Interventions: Device: MIE
- Control group (Active Comparator): Maintained following national guidelines.
  Interventions: Device: MIE

INTERVENTIONS:
Device: MIE — Two sequences separated for 1 min of 6 cycles each of MI-E(Cough Assist E70, Respironics Philips.

SUMMARY:
The main objective of the project is to determine the variation of PaO2 / FiO2 (PaFi) after the use of mechanical insufflation-exsufflation (MI-E) or mechanical cough assistant in the donor in brain death (DBD) and in the potential donor in control donor after circulatory death (cDCD) It is a randomized prospective multicentre study. Four centres with a solid organ donation program will participate in the study, the Hospital Clínic i Provincial de Barcelona (HCB), the Germans Tries y Pujol Hospital (HGTP), the Marqués de Valdecilla Hospital (HMV) and the Vall d'Hebron Hospital (HVH). One hundred and sixty consecutive eligible donors will be included in DBD and cDCD older than 18 years.

* P1: Eighty donors will be maintained following national guidelines.
* P2: Eighty donors will be maintained following national guidelines and:
* Manual techniques of secretion drainage
* Two sequences separated for 1 min of 6 cycles each of MI-E(Cough Assist E70, Respironics Philips.

Demographic variables of the donor and recipient will be collected, as well as differences in PaFi, static compliance, and radiographic changes between P1 and P2 donors. The percentage of lung donors recovered by P2 with respect to P1 will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Organ donor older than 18yo

Exclusion Criteria:

* Absolute contraindications for MIE's use
* Absolute contraindications for organ donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The changes in Oxygenation | Ten minutes after the MIE application and 60 minutes after MIE application or national protocol aplication
  The changes of oxygenation comparing MIE to national protocol

SECONDARY OUTCOMES:
Rate of complications with the use of MIE | During the intervention and 60 minutes after it.
  To analyse the complications associated with the use of MIE in organ donors
Number of potential lung donors | during the recruitment time
  To analyse the increase in potential lung donors with MIE
Number of lung donors | during the recruitment time
  To analyse the increase in lung donors with MIE

CONTACTS AND LOCATIONS:
Overall Officials: Irene bello, Professor, Study Chair — Vall d'Hebron Institute of Research
Locations (1):
- Irene bello, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: IPD will become available since the publications during 3 years
Access Criteria: IPD will be available for researchers involved in organ donation, respiratory physiotherapy or lung transplantation who asked by email to main researcher.

REFERENCES:
- [Background] Stiller K. Physiotherapy in intensive care: an updated systematic review. Chest. 2013 Sep;144(3):825-847. doi: 10.1378/chest.12-2930. PMID 23722822
- [Background] Battaglini D, Robba C, Caiffa S, Ball L, Brunetti I, Loconte M, Giacobbe DR, Vena A, Patroniti N, Bassetti M, Torres A, Rocco PR, Pelosi P. Chest physiotherapy: An important adjuvant in critically ill mechanically ventilated patients with COVID-19. Respir Physiol Neurobiol. 2020 Nov;282:103529. doi: 10.1016/j.resp.2020.103529. Epub 2020 Aug 17. PMID 32818606
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] Fernandez-Carmona A, Olivencia-Pena L, Yuste-Ossorio ME, Penas-Maldonado L; Grupo de Trabajo de Unidad de Ventilacion Mecanica Domiciliaria de Granada. Ineffective cough and mechanical mucociliary clearance techniques. Med Intensiva (Engl Ed). 2018 Jan-Feb;42(1):50-59. doi: 10.1016/j.medin.2017.05.003. Epub 2017 Jun 12. English, Spanish. PMID 28619528
- [Background] Ferreira de Camillis ML, Savi A, Goulart Rosa R, Figueiredo M, Wickert R, Borges LGA, Galant L, Teixeira C. Effects of Mechanical Insufflation-Exsufflation on Airway Mucus Clearance Among Mechanically Ventilated ICU Subjects. Respir Care. 2018 Dec;63(12):1471-1477. doi: 10.4187/respcare.06253. Epub 2018 Jul 17. PMID 30018175
- [Background] Lachal R, Louis B, Subtil F, Guerin C. Bench Assessment of the Effect of a Collapsible Tube on the Efficiency of a Mechanical Insufflation-Exsufflation Device. Respir Care. 2019 Jul;64(7):752-759. doi: 10.4187/respcare.06478. Epub 2019 Mar 12. PMID 30862688
- [Background] Morrow B, Zampoli M, van Aswegen H, Argent A. Mechanical insufflation-exsufflation for people with neuromuscular disorders. Cochrane Database Syst Rev. 2013 Dec 30;(12):CD010044. doi: 10.1002/14651858.CD010044.pub2. PMID 24374746
- [Background] Sanchez-Garcia M, Santos P, Rodriguez-Trigo G, Martinez-Sagasti F, Farina-Gonzalez T, Del Pino-Ramirez A, Cardenal-Sanchez C, Busto-Gonzalez B, Requesens-Solera M, Nieto-Cabrera M, Romero-Romero F, Nunez-Reiz A. Preliminary experience on the safety and tolerability of mechanical "insufflation-exsufflation" in subjects with artificial airway. Intensive Care Med Exp. 2018 Apr 3;6(1):8. doi: 10.1186/s40635-018-0173-6. PMID 29616357
- [Background] Bach JR. Noninvasive Respiratory Management of Patients With Neuromuscular Disease. Ann Rehabil Med. 2017 Aug;41(4):519-538. doi: 10.5535/arm.2017.41.4.519. Epub 2017 Aug 31. PMID 28971036
- [Background] Guerin C, Bourdin G, Leray V, Delannoy B, Bayle F, Germain M, Richard JC. Performance of the coughassist insufflation-exsufflation device in the presence of an endotracheal tube or tracheostomy tube: a bench study. Respir Care. 2011 Aug;56(8):1108-14. doi: 10.4187/respcare.01121. PMID 21801577
- [Background] Volpe MS, Naves JM, Ribeiro GG, Ruas G, Amato MBP. Airway Clearance With an Optimized Mechanical Insufflation-Exsufflation Maneuver. Respir Care. 2018 Oct;63(10):1214-1222. doi: 10.4187/respcare.05965. Epub 2018 Jul 17. PMID 30018177
- [Background] Bach JR, Saporito LR, Shah HR, Sinquee D. Decanulation of patients with severe respiratory muscle insufficiency: efficacy of mechanical insufflation-exsufflation. J Rehabil Med. 2014 Nov;46(10):1037-41. doi: 10.2340/16501977-1874. PMID 25096928
- [Background] Toussaint M. The use of mechanical insufflation-exsufflation via artificial airways. Respir Care. 2011 Aug;56(8):1217-9. doi: 10.4187/respcare.01448. No abstract available. PMID 21801584
- [Background] Rose L. Strategies for weaning from mechanical ventilation: a state of the art review. Intensive Crit Care Nurs. 2015 Aug;31(4):189-95. doi: 10.1016/j.iccn.2015.07.003. Epub 2015 Jul 21. PMID 26209016
- [Background] Goncalves MR, Honrado T, Winck JC, Paiva JA. Effects of mechanical insufflation-exsufflation in preventing respiratory failure after extubation: a randomized controlled trial. Crit Care. 2012 Dec 12;16(2):R48. doi: 10.1186/cc11249. PMID 22420538
- [Background] Terzi N, Prigent H, Lofaso F. Mechanical Insufflation-Exsufflation to Improve Secretion Clearance During Invasive Ventilation. Respir Care. 2018 Dec;63(12):1577-1578. doi: 10.4187/respcare.06700. No abstract available. PMID 30467229
- [Background] Nunes LC, Rizzetti DA, Neves D, Vieira FN, Kutchak FM, Wiggers GA, Pecanha FM. Mechanical insufflation/exsufflation improves respiratory mechanics in critical care: Randomized crossover trial. Respir Physiol Neurobiol. 2019 Aug;266:115-120. doi: 10.1016/j.resp.2019.05.008. Epub 2019 May 13. PMID 31096012
- [Background] Minambres E, Ballesteros MA, Rodrigo E, Garcia-Miguelez A, Llorca J, Ruiz JC, Arias M. Aggressive lung donor management increases graft procurement without increasing renal graft loss after transplantation. Clin Transplant. 2013 Jan-Feb;27(1):52-9. doi: 10.1111/j.1399-0012.2012.01690.x. Epub 2012 Aug 16. PMID 22897405
- [Background] Minambres E, Perez-Villares JM, Chico-Fernandez M, Zabalegui A, Duenas-Jurado JM, Misis M, Mosteiro F, Rodriguez-Caravaca G, Coll E. Lung donor treatment protocol in brain dead-donors: A multicenter study. J Heart Lung Transplant. 2015 Jun;34(6):773-80. doi: 10.1016/j.healun.2014.09.024. Epub 2014 Sep 28. PMID 25447580
- [Background] Benazzo A, Schwarz S, Frommlet F, Sinn K, Schweiger T, Klikovits T, Hoda AM, Moser B, Matilla JR, Renyi Vamos F, Lang G, Jaksch P, Di Nardo M, Del Sorbo L, Taghavi S, Keshavjee S, Klepetko W, Cypel M, Hoetzenecker K. Donor ventilation parameters as predictors for length of mechanical ventilation after lung transplantation: Results of a prospective multicenter study. J Heart Lung Transplant. 2021 Jan;40(1):33-41. doi: 10.1016/j.healun.2020.10.008. Epub 2020 Oct 28. PMID 33246712